CLINICAL TRIAL: NCT01145040
Title: NOMOTHETICOS: Nonlinear Modelling of Thyroid Hormones' Effect on Thyrotropin Incretion in Confirmed Open-loop Situation. A Correlation Study
Brief Title: NOMOTHETICOS: Nonlinear Modelling of Thyroid Hormones' Effect on Thyrotropin Incretion in Confirmed Open-loop Situation
Acronym: NOMOTHETICOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, PD Dr. Johannes W. Dietrich, MD, Senior consultant endocrinologist, Ruhr University of Bochum
Other Study IDs: TFC-UK10; 3718-10 (Other: Ethics commission of the Ruhr University of Bochum); U1111-1122-3273 (Registry Identifier: WHO ICTRP Universal Trial Number (UTN)); DRKS00003153 (Registry Identifier: DRKS (German Clinical Trials Register))
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hypothyroidism; Hyperthyroidism
Keywords: Overt primary hypothyroidism; Overt primary hyperthyroidism; Thyrotropic feedback control; Mathematical modelling; Nonlinear modelling; Thyroid; Pituitary; Physiological cybernetics; Full-dose levothyroxine substitution therapy; Syndrome T
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism; Thyroid Diseases; Pituitary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Partition 1: Overt primary hypothyroidism
- Partition 2: Hypothyroidism with "full dose" levothyroxine substitution therapy (more than 1.75 µg per kg of body mass)
- Partition 3: Overt primary hyperthyroidism

SUMMARY:
The NOMOTHETICOS study is a unicentric cross-sectional study for a quantitative analysis of feedback-inhibition in the thyrotropic homeostatic control. Structural parameters are obtained in vivo from open-loop analysis in patients with disconnected feedback, i.e. with overt thyroid dysfunction or full dose substitution therapy with levothyroxine.

DETAILED DESCRIPTION:
Control of thyroid hormone homeostasis is essential for function and development of the organism and hence for individual health. It is therefore not surprising that the thyroid's function is controlled by a complex, multi-loop feedback control system.

Today, the central component of the thyrotropic feedback control system is still poorly understood on a physiological level. Therefore, in mathematical models different functional relations describing the feedback-inhibition of thyrotropin incretion by thyroid hormones have been suggested [Danziger and Elmergreen 1956, Roston 1959, Norwich and Reiter 1965, DiStefano and Stear 1968, DiStefano 1969, Saratchandran et al. 1973, Li et al. 1995, Dietrich et al. 2004, Degon et al. 2008, Jonklaas and Soldin 2008, Hörmann et al. 2010]. Most of these models fail in delivering biochemical explanations for the functional interrelations they postulate.

Nevertheless, some clinical applications of these models have been developed, although their diagnostical potential is usually rather limited [Yagi et al. 1997, Pohlenz et al. 1999, Jostel et al. 2009].

Assuming that the pituitary's response to peripheral thyroid hormones is determined by active transmembrane thyroxine transport mechanisms [Dietrich et al. 2008], intracellular deiodination of thyroxine (T4), binding of resulting triiodothyronine (T3) to iodothyronine receptors and, finally, their inhibiting effect on mRNA expression, translation and release of TRH, a novel, physiologically motivated model has been developed that is based on compartment-analytical approaches, Michaelis-Menten kinetics and non competitive divisive inhibition [Dietrich et al 2004]. However, this model has not been sufficiently evaluated in a clinical context.

It is the aim of the NOMOTHETICOS study to deliver new systems-level insights into the pituitary's thyrotropic function. This unicentric cross-sectional study compares different models of feedback-inhibition by means of modern statistical methods like nonlinear regression and Akaike information criterion. Structural parameters are obtained in vivo from open-loop analysis in patients with disconnected feedback in equilibrium.

These parameters can serve as theoretical basis for possible future trials developing advanced diagnostical evaluation methods of thyrotropic pituitary function.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with disconnected feedback control due to the following conditions:

  * Overt primary hypothyroidism with TSH level higher than 10 mU/l and FT4 concentration below 7 pmol/L (5.4 ng/L) (Partition 1)
  * Overt primary hyperthyroidism with TSH level below 0.1 mU/l and FT4 concentration higher than 18 pmol/L (14 ng/L) (Partition 3)
  * All other constellations, if the patient receives substitution therapy with more 1.75 µg Levothyroxin per kg of body mass (Partition 2).
* System in equilibrium (e.g. unchanged substitution dose over the past six weeks)

Exclusion Criteria:

* Pituitary or hypothalamic dysfunction
* Severe illness that may be associated with euthyroid sick syndrome (non-thyroidal illness syndrome)
* Medication influencing pituitary function
* Pregnancy
* Missing consent for participation in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients with "open-loop" thyrotropic feedback control (disconnection at the site of the thyroid)
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Nonlinear correlation of thyrotropin levels with peripheral levothyroxine levels. | Data of individual patients are obtained one work day after consultation (to allow for laboratory investigations). Model comparison will take place immediately after the inclusion of the 100th patient.
  Nonlinear modeling of the pituitary response with different models (logarithmic, polynomial, non-competitive divisive inhibition). Selection of one out of different possible mathematical models that suffices an optimal combination of
  * best nonlinear fit (minimal p-value),
  * minimal entropy (as expressed by minimal values for Akaike information criterion, Bayesian information criterion and Hannan-Quinn information criterion) and
  * best compatibility with biochemical mechanisms.

SECONDARY OUTCOMES:
Parameters of feedback inhibition. | Data of individual patients are obtained one work day after consultation (to allow for laboratory investigations). Parameter estimation will take place immediately after the inclusion of the 100th patient.
  Extraction of structural parameters out of the model that has been selected (see primary outcome measure)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes W Dietrich, M.D., Principal Investigator — Medical Hospital I, Bergmannsheil University Hospitals, Ruhr University of Bochum; Harald H Klein, M.D., Study Chair — Medical Hospital I, Bergmannsheil University Hospitals, Ruhr University of Bochum; Johannes W Dietrich, M.D., Study Director — Medical Hospital I, Bergmannsheil University Hospitals, Ruhr University of Bochum; Bojana Bazika-Gerasch, M.D., Principal Investigator — Medical Hospital I, Bergmannsheil University Hospitals, Ruhr University of Bochum
Locations (3):
- Germany (3):
  - Klinikum Ludwigsburg-Bietigheim, Bietigheim, Baden-Wurttemberg
  - Institute for diagnostical radiology, interventional radiology and nuclear medicine, Bergmannsheil University Hospitals, Ruhr University of Bochum, Bochum, North Rhine-Westphalia
  - Medical Hospital I, Bergmannsheil University Hospitals, Ruhr University of Bochum, Bochum, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.
Supporting Information: Analytic Code

REFERENCES:
- [Background] Norwich KH, Reiter R. Homeostatic control of thyroxin concentration expressed by a set of linear differential equations. Bull Math Biophys. 1965 Jun;27(2):133-44. doi: 10.1007/BF02498768. No abstract available. PMID 5832691
- [Background] DiStefano JJ 3rd, Stear EB. Neuroendocrine control of thyroid secretion in living systems: a feedback control system model. Bull Math Biophys. 1968 Mar;30(1):3-26. doi: 10.1007/BF02476936. No abstract available. PMID 4969955
- [Background] DiStefano JJ 3rd. A model of the normal thyroid hormone glandular secretion mechanism. J Theor Biol. 1969 Mar;22(3):412-7. doi: 10.1016/0022-5193(69)90013-7. No abstract available. PMID 5803330
- [Background] Saratchandran P, Carson ER, Reeve J. An improved mathematical model of human thyroid hormone regulation. Clin Endocrinol (Oxf). 1976 Sep;5(5):473-83. doi: 10.1111/j.1365-2265.1976.tb01976.x. PMID 825330
- [Background] Li G, Liu B, Liu Y. A dynamical model of the pulsatile secretion of the hypothalamo-pituitary-thyroid axis. Biosystems. 1995;35(1):83-92. doi: 10.1016/0303-2647(94)01484-o. PMID 7772725
- [Background] Degon M, Chipkin SR, Hollot CV, Zoeller RT, Chait Y. A computational model of the human thyroid. Math Biosci. 2008 Mar;212(1):22-53. doi: 10.1016/j.mbs.2007.10.009. Epub 2007 Nov 6. PMID 18291425
- [Background] Dietrich JW, Brisseau K, Boehm BO. [Absorption, transport and bio-availability of iodothyronines]. Dtsch Med Wochenschr. 2008 Aug;133(31-32):1644-8. doi: 10.1055/s-0028-1082780. German. PMID 18651367
- [Background] Yagi H, Pohlenz J, Hayashi Y, Sakurai A, Refetoff S. Resistance to thyroid hormone caused by two mutant thyroid hormone receptors beta, R243Q and R243W, with marked impairment of function that cannot be explained by altered in vitro 3,5,3'-triiodothyroinine binding affinity. J Clin Endocrinol Metab. 1997 May;82(5):1608-14. doi: 10.1210/jcem.82.5.3945. PMID 9141558
- [Background] Pohlenz J, Weiss RE, Macchia PE, Pannain S, Lau IT, Ho H, Refetoff S. Five new families with resistance to thyroid hormone not caused by mutations in the thyroid hormone receptor beta gene. J Clin Endocrinol Metab. 1999 Nov;84(11):3919-28. doi: 10.1210/jcem.84.11.6080. PMID 10566629
- [Background] Jostel A, Ryder WD, Shalet SM. The use of thyroid function tests in the diagnosis of hypopituitarism: definition and evaluation of the TSH Index. Clin Endocrinol (Oxf). 2009 Oct;71(4):529-34. doi: 10.1111/j.1365-2265.2009.03534.x. Epub 2009 Feb 18. PMID 19226261
- [Background] Jonklaas J, Soldin SJ. Tandem mass spectrometry as a novel tool for elucidating pituitary-thyroid relationships. Thyroid. 2008 Dec;18(12):1303-11. doi: 10.1089/thy.2008.0155. PMID 19067639
- [Background] Danziger L, Elmergreen GL. The Thyroid-Pituitary Homeostatic Mechanism. Bulletin of Mathematical Biophysics 18 : 1-13, 1956.
- [Background] Roston S: Mathematical Represention of Some Endocrinological Systems. Bulletin of Mathematical Biophysics, 21:271-282, 1959.
- [Background] Dietrich JW,Tesche A, Pickardt, CR, Mitzdorf U. Thyrotropic Feedback Control: Evidence for an Additional Ultrashort Feedback Loop from Fractal Analysis. Cybernetics and Systems 35 (4): 315-31, 2004.
- [Background] Hoermann R, Eckl W, Hoermann C, Larisch R. Complex relationship between free thyroxine and TSH in the regulation of thyroid function. Eur J Endocrinol. 2010 Jun;162(6):1123-9. doi: 10.1530/EJE-10-0106. Epub 2010 Mar 18. PMID 20299491
- [Background] Dietrich JW, Landgrafe G, Fotiadou EH. TSH and Thyrotropic Agonists: Key Actors in Thyroid Homeostasis. J Thyroid Res. 2012;2012:351864. doi: 10.1155/2012/351864. Epub 2012 Dec 30. PMID 23365787
- [Background] Dietrich JW, Leow MK, Goede SL, Midgley JE, Landgrafe G, Hoermann R. Do thyroid-stimulating hormone, body weight, or body mass index serve as adequate markers to guide levothyroxine dose titration? J Am Coll Surg. 2013 Oct;217(4):752-3. doi: 10.1016/j.jamcollsurg.2013.06.008. No abstract available. PMID 24054412
- [Background] Dietrich JW, Landgrafe-Mende G, Wiora E, Chatzitomaris A, Klein HH, Midgley JE, Hoermann R. Calculated Parameters of Thyroid Homeostasis: Emerging Tools for Differential Diagnosis and Clinical Research. Front Endocrinol (Lausanne). 2016 Jun 9;7:57. doi: 10.3389/fendo.2016.00057. eCollection 2016. PMID 27375554
- [Background] Dietrich JW, Midgley JEM, Hoermann R. Editorial: "Homeostasis and Allostasis of Thyroid Function". Front Endocrinol (Lausanne). 2018 Jun 5;9:287. doi: 10.3389/fendo.2018.00287. eCollection 2018. No abstract available. PMID 29922229
- [Background] Berberich J, Dietrich JW, Hoermann R, Muller MA. Mathematical Modeling of the Pituitary-Thyroid Feedback Loop: Role of a TSH-T3-Shunt and Sensitivity Analysis. Front Endocrinol (Lausanne). 2018 Mar 21;9:91. doi: 10.3389/fendo.2018.00091. eCollection 2018. PMID 29619006